CLINICAL TRIAL: NCT01312246
Title: EnSeal Efficacy and Bursting Pressure in Human Vessels
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Prasad Leela, university of Illinois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010-0878
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Colon and Rectal Diseases
Keywords: vessel ligation; colon resection
MeSH Terms: conditions — Rectal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EnSeal Device — measurement of bursting pressure of colonic vessels after using the EnSeal Device
  Other Names: EnSeal Device- Ethicon Endo Surgery

SUMMARY:
In this study the investigators will include adult patients who are not part of a vulnerable patient population. Inclusion criteria include patients who will be undergoing resection of part of their colon that will require dividing the IMA. The investigators will use the resected surgical specimens for our project. The investigators will use the EnSeal on all major vessels in our procedure. The investigators will use the EnSeal 5 mm round head model. Due to the nature of the project, we will apply for IRB approval prior to beginning our research. The investigators plan to include 60 total patients in the study, 30 at the University of Illinois and 30 at Lutheran General Hospital.

Prior to resection, the investigators will use a sterile caliper to take an in-vivo measurement of the IMA and IMV. Immediately after resection, the investigators will remove the sealed proximal end of the IMA and the 3 cm distal to it from the surgical specimen. The investigators will similarly prepare the IMV. The investigators will inspect our vessels for any iatrogenic traumatic tears. If the vessels are suitable, the investigators will then gentle apply manual traction to remove any blood or clots within the lumen. The investigators will measure the outer diameter of the vessels using a digital caliper. If there are small branches, the investigators will tie them off with suture. The unsealed end will then be attached to the burst pressure tester with suture and it will be tested for the bursting pressure. The device measures pressure continuously as it infuses the segment with normal saline at a steady rate (50 ml/hr). A leak will be determined by a decrease in intra-luminal pressure of 100 mm Hg or a visible leak. A failure to seal the vessels will be determined by a bursting pressure of less than 100 mm Hg. It should be noted that each section would only be pressure-tested once. All of our data will be collected on the enclosed data sheet we have created for use in this protocol. The investigators will then place the vessels with the original surgical specimen where it will be submitted for routine pathological examination of surgical specimens. Twenty five specimens at each site will undergo the testing, whereas 5 specimens will be sent to pathology without testing.

Our pathologist will analyze the submitted specimen for extent of seal, disruption of vessel smooth muscle, gas bubbles, and will stain for elastin to analyze the disruption in the vessel wall. In addition, the seal will be measured and we will obtain digital images. The specimens submitted for pathology will be 5 burst specimens as well as 5 un-burst specimens taken from the pool of 25 patients at UIC.

For our human component, the investigators have estimated the standard deviation and width of the confidence interval to be 100 mm Hg each. With a 95% confidence level, the investigators expect to require 16 measurements for human specimens from 16 patients although the investigators will use 50 patients to allow for errors in obtaining pressures.

Our timeline for the completion of the projects is 6 months. The investigators plan on being able to complete the human burst pressure testing within 6 months.

DETAILED DESCRIPTION:
Introduction

Multiple new cautery devices are used to perform quicker and safer surgeries. These devices are able to seal vessels without need of ties or adjunct maneuvers and produce a minimal thermal spread to adjacent tissues. We have found that the EnSeal is a reliable, versatile, and effective device for sealing vessels.

Currently, the EnSeal is approved for vessels as large as 7 mm in diameter. We believe, based on prior clinical experience, that the EnSeal can safely seal vessels of a larger diameter. Current data shows that the bursting pressures obtained in 7 mm vessels are five times the physiological normal pressure in animal models.1, 2 We have demonstrated that all of the mesenteric vessels encountered in a human colectomy can be safely divided with EnSeal. However, neither we nor other researchers have measured the bursting pressure of these seals in human patients.

We propose to examine the bursting pressures of vessels taken in colectomies in an ex-vivo fashion. After we use the EnSeal to divide the inferior mesenteric artery at its origin, we will then use assess the bursting pressure of this seal. We will similarly assess the inferior mesenteric vein. We will measure the diameter of the vessels both in-vivo and ex-vivo. Finally, we will conduct histopathological examination of the sealed vessels to determine the effects of the EnSeal device on the structure of the vessels.

Background

With the increased preference for laparoscopic surgery, new instruments are needed to safely replicate and, where possible, improve upon the techniques used in open surgery. Visualization is eminently important and dependent on multiple factors, including bleeding and smoke from coagulation and cautery. Therefore, there is a high demand for devices that can safely coagulate tissue with low heat and little smoke. Resection of tissues in a safe and haemostatic fashion in laparoscopic colorectal surgery depends upon good control of mesenteric vessels. Ideally, the thermal spread should be minimal and travel in a predictable pattern. Various new devices have been created and used for the purposes of vessel sealing, with some of the more popular being Ligasure (Valleylab), Harmonic (Ethicon), Gyrus (Gyrus ACMI), and EnSeal (Ethicon). Multi-purpose instruments are preferable because the surgeon can avoid frequent exchange of instruments and thus reduce operative time. The previously mentioned vessel-sealing devices work with two jaws and can also be used to manipulate some tissue. Of particular interest to our group of colorectal surgeons is the finding that along with decreased operative time, these devices have been shown to contribute to decreased blood loss during laparoscopic colectomies.3 These modern vessel-sealing devices work by varying methods. The Harmonic Scalpel is an ultrasonic shear that breaks hydrogen bonds and cause tissue coagulation and vessel sealing.4 The Ligasure device works by coagulating the tissue in the jaws of the device with high-current/low-voltage flow and then using high-pressure jaws to seal it.5 The nano-particle technology of the EnSeal device aims to lower the temperature of the instrument to minimize heat transfer to adjacent tissue and allows for different temperatures within different parts of the jaws. It turns off when collagen denatures, at approximately 100 degrees Celsius.6 These sealing systems have been widely used in many surgical disciplines and surgeons continue to try to find new uses for these innovative devices. They have been compared to conventional methods such as clips and ties and found to be as effective when applied properly.7 The Gyrus PK system has been used in urological and robotic surgery.8, 9 The Harmonic Scalpel has been used in major abdominal operations and also in otolaryngology operations.10, 11 Ligasure has perhaps been the most widely adopted and is used in gynecological, otolaryngology, and colorectal specialties.12-15 The EnSeal device is newer than the others and while it is gaining popularity in its use, it has not been as extensively studied at this time.

Currently, the USA FDA has approved the EnSeal device for vessels up to 7 mm in diameter. This is equal or greater to other vessel sealing systems that are widely used such as Ligasure (7 mm) and Harmonic Scalpel (5 mm). Porcine studies done by SurgRx as well as research groups from Cleveland Clinic - FL and Carolinas Medical Center demonstrate the safety of this device in its approved size range when compared to other devices. In these studies, they find that the EnSeal has significantly higher burst pressures on sealed vessels than other sealing systems (678 mm Hg for EnSeal vs 489 mm Hg for Ligasure) or that there is no statistical difference, but that it seals at supra-physiologic pressures (891 mm Hg EnSeal vs 884 mm Hg Ligasure).1, 2 These measurements are obtained by securing the open end of a vessel to a device that fills the lumen with fluid. Once the seal on the other end bursts, the machine records the final pressure reading within the lumen of the vessel. Other notable findings of the EnSeal include less adventitial damage to the vessels on histopathologic evaluation and minimal failure rates (only 1/39 vessels failed to seal).1, 2 A study completed from Turkey used EnSeal on rat liver parenchyma and compared it to Ligasure and conventional methods for liver resection. Sahin and colleagues found that EnSeal was at least as effective as conventional techniques and that there was less inflammation and damage due to thermal spread to the rat liver parenchyma when compared to Ligasure.16 In a comparison of two ultrasonic devices on human vessels, Ching found that veins have a decreasing burst pressure as the diameter of the vessels increase.17 These burst pressures are much lower than what is reported in porcine arteries. This finding makes it important to determine the seal bursting pressure in human vessels so that the relationship between experimental values in porcine models can be clinically correlated. Previous studies have analyzed the histopathologic effect of the EnSeal device on the blood vessels.2 We will also do an analysis of human tissue.

In our practice, we routinely use the EnSeal device to seal the ileocolic vessels and the inferior mesenteric artery and vein (IMA, IMV). Data with good evidence of the diameter (external or internal) of the inferior mesenteric artery is not widely available. However, we were able to find some data that can provide a little information. In a study by Yekeler et al, the investigators used ultrasound technology to determine the internal diameter of the superior mesenteric artery (SMA). In their study, they found that in healthy patients the internal diameter average was 5.8 mm. Among their findings is a pattern of significantly increased internal diameter in patients with active inflammation compared to patients with quiescent disease.18 We have long suspected that in tissue experiencing acute or chronic inflammation the feeding vessel will be larger; their evidence supports this hypothesis. In a very small study examining the use of the IMA for coronary artery bypass grafts, researchers harvested two IMAs and measured one of them. This artery had a 4 mm diameter at its origin. The IMA is smaller than the SMA in the vast majority of patients. Therefore, the findings by Shatapathy are consistent with this expectation.19 In our practice, we have gravitated towards the EnSeal. We find that it is effective, reliable and its versatility is evidenced by its use as a grasper, dissector, scissors and vessel and soft-tissue sealer. The nano-particles that are within the jaws of the device to regulate current and heat distribution serve to protect the adjacent tissue from thermal injury. Such injuries from other devices have been documented and often present with late and serious complications.21 As part of our normal surgical practice, we use the EnSeal to divide and seal the inferior mesenteric artery and vein when their resection is indicated. In our experience with this device, it has a low failure rate. We have not experienced any post-operative bleeding that requires transfusion or re-operation. Even though we believe that the majority of IMAs we encounter are below the 7 mm size, most surgeons do not feel comfortable using the EnSeal to seal this vessel and will use staplers to divide them.

We intend to demonstrate that the bursting pressures in large vessels (IMA, IMV) sealed in colectomy of human patients are sufficiently high. Using the EnSeal device on larger vessels, we believe, would further reduce operating time, blood loss, and hasten post-operative recovery from less tissue manipulation.

Methods

In this study we will include adult patients who are not part of a vulnerable patient population. Inclusion criteria include patients who will be undergoing resection of part of their colon that will require dividing the IMA. We will use the resected surgical specimens for our project. We will use the EnSeal on all major vessels in our procedure. We will use the EnSeal 5 mm round head model. Due to the nature of the project, we will apply for IRB approval prior to beginning our research. We plan to include 60 total patients in the study, 30 at the University of Illinois and 30 at Lutheran General Hospital.

Prior to resection, we will use a sterile caliper to take an in-vivo measurement of the IMA and IMV. Immediately after resection, we will remove the sealed proximal end of the IMA and the 3 cm distal to it from the surgical specimen. We will similarly prepare the IMV. We will inspect our vessels for any iatrogenic traumatic tears. If the vessels are suitable, we will then gentle apply manual traction to remove any blood or clots within the lumen. We will measure the outer diameter of the vessels using a digital caliper. If there are small branches, we will tie them off with suture. The unsealed end will then be attached to the burst pressure tester with suture and it will be tested for the bursting pressure. The device measures pressure continuously as it infuses the segment with normal saline at a steady rate (50 ml/hr). A leak will be determined by a decrease in intra-luminal pressure of 100 mm Hg or a visible leak. A failure to seal the vessels will be determined by a bursting pressure of less than 100 mm Hg. It should be noted that each section would only be pressure-tested once. All of our data will be collected on the enclosed data sheet we have created for use in this protocol. We will then place the vessels with the original surgical specimen where it will be submitted for routine pathological examination of surgical specimens. Twenty five specimens at each site will undergo the testing, whereas 5 specimens will be sent to pathology without testing.

Our pathologist will analyze the submitted specimen for extent of seal, disruption of vessel smooth muscle, gas bubbles, and will stain for elastin to analyze the disruption in the vessel wall. In addition, the seal will be measured and we will obtain digital images. The specimens submitted for pathology will be 5 burst specimens as well as 5 un-burst specimens taken from the pool of 25 patients at UIC.

For our human component, we have estimated the standard deviation and width of the confidence interval to be 100 mm Hg each. With a 95% confidence level, we expect to require 16 measurements for human specimens from 16 patients although we will use 50 patients to allow for errors in obtaining pressures.

Our timeline for the completion of the projects is 6 months. We plan on being able to complete the human burst pressure testing within 6 months.

Budget

The budget PAF number has been included in this study. The budget also includes moneys for a concurrent study involving porcine vessels. We will harvest these blood vessels after pigs used for other research purposes are euthanized. I have included a letter from the BRL stating that this study does not require approval because we are using animals that were used for other purposes.

ELIGIBILITY:
Inclusion Criteria:

* Include patients who will be undergoing resection of part of their colon that will require dividing the colonic vessels. The use of the resected surgical specimens is included our project.

Exclusion Criteria:

* Patients who do not meet the the inclusion criteria.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
EnSeal Efficacy and Bursting Pressures in Human Vessels | 21 months
  Demonstrate that the bursting pressures in large vessels (IMA, IMV) sealed in colectomy of human patients are sufficiently high. Using the EnSeal device on larger vessels, the investigators believe, would further reduce operating time, blood loss, and hasten post-operative recovery from less tissue manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Leela M Prasad, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University Of Illinois Medical Center at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Newcomb WL, Hope WW, Schmelzer TM, Heath JJ, Norton HJ, Lincourt AE, Heniford BT, Iannitti DA. Comparison of blood vessel sealing among new electrosurgical and ultrasonic devices. Surg Endosc. 2009 Jan;23(1):90-6. doi: 10.1007/s00464-008-9932-x. Epub 2008 May 16. PMID 18483824
- [Background] Person B, Vivas DA, Ruiz D, Talcott M, Coad JE, Wexner SD. Comparison of four energy-based vascular sealing and cutting instruments: A porcine model. Surg Endosc. 2008 Feb;22(2):534-8. doi: 10.1007/s00464-007-9619-8. Epub 2007 Dec 20. PMID 18097720
- [Background] Campagnacci R, de Sanctis A, Baldarelli M, Rimini M, Lezoche G, Guerrieri M. Electrothermal bipolar vessel sealing device vs. ultrasonic coagulating shears in laparoscopic colectomies: a comparative study. Surg Endosc. 2007 Sep;21(9):1526-31. doi: 10.1007/s00464-006-9143-2. Epub 2007 Feb 8. PMID 17287913
- [Background] Entezari K, Hoffmann P, Goris M, Peltier A, Van Velthoven R. A review of currently available vessel sealing systems. Minim Invasive Ther Allied Technol. 2007;16(1):52-7. doi: 10.1080/13645700601181414. PMID 17365677
- [Background] Gilleran JP, Thaly RK, Chernoff AM. Rapid communication: bipolar PlasmaKinetic transurethral resection of the prostate: reliable training vehicle for today's urology residents. J Endourol. 2006 Sep;20(9):683-7. doi: 10.1089/end.2006.20.683. PMID 16999627
- [Background] Meehan JJ. The robotic Gyrus PK: a new articulating thermal sealing device and a preliminary series report. J Laparoendosc Adv Surg Tech A. 2008 Feb;18(1):183-5. doi: 10.1089/lap.2007.0179. PMID 18266601
- [Background] Kang SK, Kunanandam T, Clark L. Prospective, case-control study of surgical efficiency of ultrasonic shear ('harmonic scalpel') thyroidectomy compared with conventional thyroidectomy. J Laryngol Otol. 2008 Nov;122(11):1194-6. doi: 10.1017/S0022215107001661. Epub 2008 Feb 19. PMID 18282338
- [Background] Lachanas VA, Hajiioannou JK, Karatzias GT, Filios D, Koutsias S, Mourgelas C. Comparison of LigaSure vessel sealing system, harmonic scalpel, and cold knife tonsillectomy. Otolaryngol Head Neck Surg. 2007 Sep;137(3):385-9. doi: 10.1016/j.otohns.2007.05.012. PMID 17765762
- [Background] Hagen B, Eriksson N, Sundset M. Randomised controlled trial of LigaSure versus conventional suture ligature for abdominal hysterectomy. BJOG. 2005 Jul;112(7):968-70. doi: 10.1111/j.1471-0528.2005.00561.x. PMID 15958001
- [Background] Hefni MA, Bhaumik J, El-Toukhy T, Kho P, Wong I, Abdel-Razik T, Davies AE. Safety and efficacy of using the LigaSure vessel sealing system for securing the pedicles in vaginal hysterectomy: randomised controlled trial. BJOG. 2005 Mar;112(3):329-33. doi: 10.1111/j.1471-0528.2004.00325.x. PMID 15713149
- [Background] Kaplan B, Wang Z, Keilani T, Kaufman DB. The specificity of monoclonal fluorescence polarization immunoassay for cyclosporine in recipients of simultaneous pancreas-kidney transplants. Ther Drug Monit. 1995 Oct;17(5):499-503. doi: 10.1097/00007691-199510000-00010. PMID 8585113
- [Background] Kossi J, Luostarinen M, Kontula I, Laato M. Laparoscopic sigmoid and rectal resection using an electrothermal bipolar vessel sealing device. J Laparoendosc Adv Surg Tech A. 2007 Dec;17(6):719-22. doi: 10.1089/lap.2006.0238. PMID 18158799
- [Background] Sahin DA, Kusaslan R, Sahin O, Akbulut G, Bas O, Dilek ON. Histopathological effects of bipolar vessel sealing devices on liver parenchyma and comparison with suture method: an experimental study. Eur Surg Res. 2007;39(2):111-7. doi: 10.1159/000099599. Epub 2007 Feb 13. PMID 17299268
- [Background] Ching SS, Verbeke CS, Homer-Vanniasinkam S, McMahon MJ. Comparison of torsional and linear mode ultrasonic coagulating shears for sealing veins. J Laparoendosc Adv Surg Tech A. 2008 Dec;18(6):819-24. doi: 10.1089/lap.2008.0066. PMID 19105669
- [Background] Yekeler E, Danalioglu A, Movasseghi B, Yilmaz S, Karaca C, Kaymakoglu S, Acunas B. Crohn disease activity evaluated by Doppler ultrasonography of the superior mesenteric artery and the affected small-bowel segments. J Ultrasound Med. 2005 Jan;24(1):59-65. doi: 10.7863/jum.2005.24.1.59. PMID 15615929
- [Background] Shatapathy P, Aggarwal BK, Punnen J. Inferior mesenteric artery as a free arterial conduit for myocardial revascularization. J Thorac Cardiovasc Surg. 1997 Jan;113(1):210-1. doi: 10.1016/S0022-5223(97)70417-3. No abstract available. PMID 9011692
- [Background] van Andel CJ, Pistecky PV, Borst C. Mechanical properties of porcine and human arteries: implications for coronary anastomotic connectors. Ann Thorac Surg. 2003 Jul;76(1):58-64; discussion 64-5. doi: 10.1016/s0003-4975(03)00263-7. PMID 12842513